CLINICAL TRIAL: NCT05430282
Title: Effect of Cervical Exercises in Addition to Vestibular Rehabilitation in the Treatment of Peripheral Vestibular Disorders
Brief Title: Cervical Exercise in Peripheral Vestibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Principal investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-9.1Y/54
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Vestibular Disorder; Peripheral Vestibular Disorder
Keywords: vestibular disorders; cervical exercises; vertigo; vestibular exercises
MeSH Terms: conditions — Vestibular Diseases; Vertigo

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator responsible for clinical assessment will be blinded to subject's intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular rehabilitation (Active Comparator): Patients in the vestibular rehabilitation group will be asked to do vestibular exercises 3 times a day for 20 minutes, every day for one month.
  Interventions: Other: Only vestibular rehabilitation; Other: Cervical exercises in addition to vestibular rehabilitation
- Cervical exercise in addition to vestibular rehabilitation (Experimental): Patients in this group will receive the same vestibular exercise program and will be asked to do additional neck exercises and they will be asked to do these exercises twice a day for ten minutes.
  Interventions: Other: Cervical exercises in addition to vestibular rehabilitation

INTERVENTIONS:
Other: Only vestibular rehabilitation — Vestibular adaptation exercises, static and dynamic balance exercises, proprioceptive and conditioning exercises.
  Arms: Vestibular rehabilitation
Other: Cervical exercises in addition to vestibular rehabilitation — Cervical range of motion exercises, stretching exercises for the trapezius muscle, isometric and isotonic strengthening exercises in addition to conventional vestibular rehabilitation exercises.

SUMMARY:
70 patients with peripheral vestibular disorders will be included in the study. Half of the subjects will receive vestibular rehabilitation exercises and the other half will receive additional cervical exercises. Results from the two groups will be compared.

DETAILED DESCRIPTION:
70 patients with a diagnosis of peripheral vestibular disease will be enrolled in the study. Patient selection will be carried out in the physiatry, otorhinolaryngology and neurology outpatient clinics of our university hospital. Eligible patients will be informed about the study and those that accept to take part in the study will be referred to an investigator for history taking and physical examination. Demographic data, medical history and examination findings will be recorded. After initial assessment, all patients will receive a short education regarding vestibular exercises that they will be asked to do at home. A second investigator will be responsible for the randomization of subjects into two groups according to a computer generated randomization table and that same investigator will prescribe the second group additional cervical exercises to do in addition to the vestibular rehabilitation exercises.

After one months, patients will be reassessed and their measurements will be recorded. Statistical analyses will be carried out to compare the outcome scores of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of peripheral vestibular disease
* Being older than 18 years of age

Exclusion Criteria:

* Psychostimulant or psychotropic drug use that might alter vestibular functions
* Severe neurological, psychiatric or orthopedic disorder that might alter patients' ability to comply with the exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline The activities-specific balance confidence (ABC) scale at 4 weeks | Baseline and 4th week visit
  A questionnaire that measures an individual's confidence during ambulatory activities. The scale is scored from 0 to 100. 100 indicates better outcome.
Change from baseline Dizziness handicap inventory at 4 weeks | Baseline and 4th week visit
  A 25-item self-report questionnaire that quantifies the impact of dizziness on daily life by measuring self-perceived handicap. The scale is scored from 0 to 100. 100 indicates better outcome.
Change from baseline Gait speed at 4 weeks | Baseline and 4th week visit
  Gait speed is the time one takes to walk a specified distance on level surfaces over a short distance. Gait speed has different reference values according to age and sex.
Change from baseline Dynamic gait index at 4 weeks | Baseline and 4th week visit
  An inventory that assesses individual's ability to modify balance while walking in the presence of external demands. Highest possible score is 24 points and lower scores indicate worse outcome.
Change from baseline Functional gait assessment at 4 weeks | Baseline and 4th week visit
  An index that is used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. Highest score is 30 points and higher scores denote better outcome.
Change from baseline Romberg test at 4 weeks | Baseline and 4th week visit
  A balance test that challenges the vestibular, proprioceptive and visual systems. Subject is asked to stand erect with eyes open/closed, on a hard/smooth surface and with feet side by side/ in tandem.Normally a person is expected to be able to stand in these positions for 30 seconds.

SECONDARY OUTCOMES:
Change from baseline Visual analog scale for neck pain at 4 weeks | Baseline and 4th week visit
  Patient reported level of neck pain on a scale from 0 to 10 centimeters. 10 denotes severe pain and 0 denotes lack of pain.
Change from baseline Visual analog scale for dizziness at 4 weeks | Baseline and 4th week visit
  Patient reported level of dizziness on a scale from 0 to 10 centimeters. 10 indicates severe dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Kirazli, Prof, Study Chair — Ege University School of Medicine
Locations (1):
- Ege University School of Medicine, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sulway S, Whitney SL. Advances in Vestibular Rehabilitation. Adv Otorhinolaryngol. 2019;82:164-169. doi: 10.1159/000490285. Epub 2019 Jan 15. PMID 30947180
- [Background] Dunlap PM, Holmberg JM, Whitney SL. Vestibular rehabilitation: advances in peripheral and central vestibular disorders. Curr Opin Neurol. 2019 Feb;32(1):137-144. doi: 10.1097/WCO.0000000000000632. PMID 30461465